CLINICAL TRIAL: NCT03621098
Title: EMPOWER-PULM (PULMonary Outcomes in Older Adults Empowered With Movement to Prevent Obesity and Weight Regain)
Acronym: EMPOWER-PULM
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00041663
Record Dates: First submitted 2018-08-01; First posted 2018-08-08 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Obesity; Pulmonary Disease; Dyspnea
Keywords: Exercise
MeSH Terms: conditions — Obesity; Lung Diseases; Dyspnea; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diet+Exercise: Diet with structured exercise (mostly walking) at a moderate-intensity level This is not an intervention study, however, the intervention type from the parent study (EMPOWER) was behavioral (Caloric Restriction with and without Structured Exercise or Daily Activity)
- Diet+Daily Activity: Diet with increased light-intensity physical activity and decreased sedentary behavior throughout the day.
  This is not an intervention study, however, the intervention type from the parent study (EMPOWER) was behavioral (Caloric Restriction with and without Structured Exercise or Daily Activity)
- Diet+Exercise+Daily Activity: Diet with structured exercise and increased daily activity. This is not an intervention study, however, the intervention type from the parent study (EMPOWER) was behavioral (Caloric Restriction with and without Structured Exercise or Daily Activity)

SUMMARY:
The purpose of this study is to improve the understanding of the effects of weight loss on the lungs in older adults. Different types of tests to understand the effects of the EMPOWER interventions on lung function will be administered.

DETAILED DESCRIPTION:
This is a randomized clinical trial of the effects of structured aerobic exercise and a sedentary behavior intervention during weight loss on respiratory function. Site will enroll 150 older (65-85 years), obese (BMI=30-45 kg/m2), sedentary men and women from EMPOWER. EMPOWER is a 3-group design where participants will undergo a 9-month weight loss (WL) intervention (6-mo intensive phase and 3-mo reduced contact phase), followed by a 9-month self-managed follow-up phase with minimal contact. The diet element of the interventions is identical across groups, but groups differ by activity intervention: 1) moderate-intensity aerobic exercise (WL+EX); 2) intervening on SB (WL+SitLess); or 3) (WL+EX+SitLess)

ELIGIBILITY:
Inclusion Criteria:

* 65 -85 years of age
* BMI = 30-45 kg/m2
* Weight stable - no loss or gain (±5%) in past 6 months
* Sedentary
* No contraindication for safe and optimal participation in exercise training
* Approved for participation by Medical Director

Exclusion Criteria:

* Dependent on cane or walker
* Reported unintentional or intentional weight loss or gain of >5% in past 6 months
* Participation in regular resistance training and/or > 20 mins/day of aerobic exercise in past 6 months
* Osteroporosis (t-score <2.3 on hip or spine scan); Severe arthritis, or other musculoskeletal disorder; Joint replacement or other orthopedic surgery in past 6 mos; joint replacement or other orthopedic surgery planned in next 2 years
* Uncontrolled resting hypertension (>160/90 mmHg);
* Current or recent past (within 1 year) severe symptomatic heart disease, uncontrolled angina, stroke, chronic respiratory disease other than asthma or COPD, any disease requiring oxygen use, neurological or hematological disease,; cancer requiring treatment in past year, except non-melanoma skin cancers
* Serious conduction disorder, new Q waves or ST-segment depression (>3mm), or uncontrolled arrhythmia
* Room air SpO2 (oxygen saturation) at rest or with exercise qualifying for supplementary oxygen (SpO2≤88%)
* Abnormal kidney or liver function (2x upper limit of normal);
* eFGR < mL/min/1.73m2
* Anemia (Hb<14 g/dl in men/<12.3 g/dL in women);
* Uncontrolled diabetes (fasting blood glucose > 140 mg/dl);
* Deficient levels of vitamin D (25 hydroxyvitamin D level <20mg/mL) in those not taking a vitamin D supplement
* Smoker (No nicotine in past yr)
* No heavy alcohol use (>14 drinks/week)
* Unstable severe depression
* Regular use of: growth hormones, oral steroids, weight loss medications* or prescription osteoporosis medications*
* Current participation in other research study

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Current participants in the parent study, EMPOWER (Empowered with Movement to Prevent Obesity and Weight Regain)
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Number of patients who are able to undergo Pulmonary Function | Month 6 (end of study)
  Number of patients who are able to undergo Pulmonary Function
Number of patients who are able to undergo respiratory muscle strength testing | Month 6 (end of study)
  Number of patients who are able to undergo respiratory muscle strength testing
Participant retention | Month 6 (end of study)
  Measured by the number of participants who return for the 6 month testing
Assess FEV1 on pulmonary function testing for breathlessness | Month 6 (end of study)
  FEV1 used to estimate treatment effect sizes on pulmonary function and physical performance.. Paired t-test analysis will be used to compare within treatment group pre-and post outcomes with adjusted analysis. ANOVA with adjusted analysis will be used to amke between group comparisons and to compare changes in outcomes between treatment groups after the 6-month intensive weight loss phase.
Assess FVC on pulmonary function testing for breathlessness | Month 6 (end of study)
  FVC used to estimate treatment effect sizes on pulmonary function and physical performance. Paired t-test analysis will be used to compare within treatment group pre- and post outcomes with adjusted analysis. ANOVA with adjusted analysis will be used to make between group comparisons and to compare changes in outcomes between treatment groups after the 6-month intensive weight loss phase.
Lung volumes | Month 6 (end of study)
  Lung volumes measures measures the volume of gas within the lungs and is considered a standard for lung volume measurements. Participants are asked to sit comfortably. They are then asked to breath through a mouthpiece that is connected to a sensor that will be recording changes in the concentration of gas washed out from the lungs with each breath taken. Scores based on mMRC (Modified Medical Research Council) dyspnea scale
Diffusing capacity | Month 6 (end of study)
  Diffusing Capacity will be measured by carbon-monoxide single-breath wash out. This test examines the alveolar uptake efficiency for carbon monoxide and therefore reflects the quality of alveolar-capillary gas uptake (how well gas diffuses through alveoli into the capillaries to get to the red blood cells).
Respiratory muscle strength | Month 6 (end of study)
  Respiratory muscle strength is assessed by measuring the maximal inspiratory the maximal expiratory pressures. The maximal inspiratory pressure reflects diaphragmatic and inspiratory muscle strength while the maximal expiratory pressure reflects abdominal muscle and expiratory muscle strength. Paired t-test analysis will be used to compare within treatment group pre- and post outcomes with adjusted analysis. ANOVA with adjusted analysis will be used to make between group comparisons and to compare changes in outcomes between treatment groups after the 6-month intensive weight loss phase.
Six minute walk distance | Month 6 (end of study)
  The 6-minute walk test s a validated test in chronic respiratory disease. It is self-paced of walking capacity and participants are encouraged to cover as much distance as they can in within 6 minutes. The 6-minute walk distance will be measured which is strongly associated with clinical outcomes. Pulse oximetry will be continuously measured
Dyspnea scores based on mMRC (Modified Medical Research Council) | Month 6 (end of study)
  The mMRC is a 1 question, five-item instrument to assess a patient's degree of breathlessness in relation to physical activity. Participants are given a brief description of an activity and then are asked to select the statement that best describes their experience with dyspnea. The score on the mMRC is weighted on a 0-4 scale and quantifies disability and exercise limitation associated with breathlessness.
Dyspnea scores based on USCD SOBQ (University of California Shortness of Breath Questionnaire) | Month 6 (end of study)
  SOBQ is a 24-item questionnaire; 21 items assess severity of breathlessness during specific activities of daily living and 3 items assess limitations due to shortness of breath, fear of harm from overexertion, and fear of shortness of breath. Each item is weighted on a 0-5 scale, and are totaled for a final score of 0-120 with high scores indicating increased severity with performing activities.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Nicklas, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lazarus R, Sparrow D, Weiss ST. Effects of obesity and fat distribution on ventilatory function: the normative aging study. Chest. 1997 Apr;111(4):891-8. doi: 10.1378/chest.111.4.891. PMID 9106566
- [Background] Jones RL, Nzekwu MM. The effects of body mass index on lung volumes. Chest. 2006 Sep;130(3):827-33. doi: 10.1378/chest.130.3.827. PMID 16963682
- [Background] Babb TG, Ranasinghe KG, Comeau LA, Semon TL, Schwartz B. Dyspnea on exertion in obese women: association with an increased oxygen cost of breathing. Am J Respir Crit Care Med. 2008 Jul 15;178(2):116-23. doi: 10.1164/rccm.200706-875OC. Epub 2008 Apr 17. PMID 18420968
- [Background] Salome CM, Munoz PA, Berend N, Thorpe CW, Schachter LM, King GG. Effect of obesity on breathlessness and airway responsiveness to methacholine in non-asthmatic subjects. Int J Obes (Lond). 2008 Mar;32(3):502-9. doi: 10.1038/sj.ijo.0803752. Epub 2007 Oct 23. PMID 17955030
- [Background] Sharma G, Goodwin J. Effect of aging on respiratory system physiology and immunology. Clin Interv Aging. 2006;1(3):253-60. doi: 10.2147/ciia.2006.1.3.253. PMID 18046878
- [Background] Rossi A, Fantin F, Di Francesco V, Guariento S, Giuliano K, Fontana G, Micciolo R, Solerte SB, Bosello O, Zamboni M. Body composition and pulmonary function in the elderly: a 7-year longitudinal study. Int J Obes (Lond). 2008 Sep;32(9):1423-30. doi: 10.1038/ijo.2008.103. Epub 2008 Jul 22. PMID 18645577
- [Background] Rossi AP, Watson NL, Newman AB, Harris TB, Kritchevsky SB, Bauer DC, Satterfield S, Goodpaster BH, Zamboni M. Effects of body composition and adipose tissue distribution on respiratory function in elderly men and women: the health, aging, and body composition study. J Gerontol A Biol Sci Med Sci. 2011 Jul;66(7):801-8. doi: 10.1093/gerona/glr059. Epub 2011 Apr 15. PMID 21498841
- [Background] Alley DE, Chang VW. The changing relationship of obesity and disability, 1988-2004. JAMA. 2007 Nov 7;298(17):2020-7. doi: 10.1001/jama.298.17.2020. PMID 17986695
- [Background] Vasquez E, Batsis JA, Germain CM, Shaw BA. Impact of obesity and physical activity on functional outcomes in the elderly: data from NHANES 2005-2010. J Aging Health. 2014 Sep;26(6):1032-46. doi: 10.1177/0898264314535635. Epub 2014 Jun 9. PMID 24913317
- [Background] American College of Cardiology/American Heart Association Task Force on Practice Guidelines, Obesity Expert Panel, 2013. Executive summary: Guidelines (2013) for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Obesity Society published by the Obesity Society and American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Based on a systematic review from the The Obesity Expert Panel, 2013. Obesity (Silver Spring). 2014 Jul;22 Suppl 2:S5-39. doi: 10.1002/oby.20821. No abstract available. PMID 24961825
- [Background] Wei YF, Tseng WK, Huang CK, Tai CM, Hsuan CF, Wu HD. Surgically induced weight loss, including reduction in waist circumference, is associated with improved pulmonary function in obese patients. Surg Obes Relat Dis. 2011 Sep-Oct;7(5):599-604. doi: 10.1016/j.soard.2011.04.221. Epub 2011 Apr 19. PMID 21689991
- [Background] Karason K, Lindroos AK, Stenlof K, Sjostrom L. Relief of cardiorespiratory symptoms and increased physical activity after surgically induced weight loss: results from the Swedish Obese Subjects study. Arch Intern Med. 2000 Jun 26;160(12):1797-802. doi: 10.1001/archinte.160.12.1797. PMID 10871973
- [Background] Babb TG, Wyrick BL, Chase PJ, DeLorey DS, Rodder SG, Feng MY, Ranasinghe KG. Weight loss via diet and exercise improves exercise breathing mechanics in obese men. Chest. 2011 Aug;140(2):454-460. doi: 10.1378/chest.10-1088. Epub 2011 Jan 27. PMID 21273293
- [Background] Held M, Mittnacht M, Kolb M, Karl S, Jany B. Pulmonary and cardiac function in asymptomatic obese subjects and changes following a structured weight reduction program: a prospective observational study. PLoS One. 2014 Sep 18;9(9):e107480. doi: 10.1371/journal.pone.0107480. eCollection 2014. PMID 25233078
- [Background] Bhammar DM, Stickford JL, Bernhardt V, Babb TG. Effect of weight loss on operational lung volumes and oxygen cost of breathing in obese women. Int J Obes (Lond). 2016 Jun;40(6):998-1004. doi: 10.1038/ijo.2016.21. Epub 2016 Feb 12. PMID 26869243
- [Background] Womack CJ, Harris DL, Katzel LI, Hagberg JM, Bleecker ER, Goldberg AP. Weight loss, not aerobic exercise, improves pulmonary function in older obese men. J Gerontol A Biol Sci Med Sci. 2000 Aug;55(8):M453-7. doi: 10.1093/gerona/55.8.m453. PMID 10952368
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Wanger J, Clausen JL, Coates A, Pedersen OF, Brusasco V, Burgos F, Casaburi R, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson D, Macintyre N, McKay R, Miller MR, Navajas D, Pellegrino R, Viegi G. Standardisation of the measurement of lung volumes. Eur Respir J. 2005 Sep;26(3):511-22. doi: 10.1183/09031936.05.00035005. No abstract available. PMID 16135736
- [Background] Macintyre N, Crapo RO, Viegi G, Johnson DC, van der Grinten CP, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, Gustafsson P, Hankinson J, Jensen R, McKay R, Miller MR, Navajas D, Pedersen OF, Pellegrino R, Wanger J. Standardisation of the single-breath determination of carbon monoxide uptake in the lung. Eur Respir J. 2005 Oct;26(4):720-35. doi: 10.1183/09031936.05.00034905. No abstract available. PMID 16204605
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Tashkin DP, Altose MD, Connett JE, Kanner RE, Lee WW, Wise RA. Methacholine reactivity predicts changes in lung function over time in smokers with early chronic obstructive pulmonary disease. The Lung Health Study Research Group. Am J Respir Crit Care Med. 1996 Jun;153(6 Pt 1):1802-11. doi: 10.1164/ajrccm.153.6.8665038.
- [Background] Colak Y, Afzal S, Lange P, Nordestgaard BG. Obese individuals experience wheezing without asthma but not asthma without wheezing: a Mendelian randomisation study of 85,437 adults from the Copenhagen General Population Study. Thorax. 2016 Mar;71(3):247-54. doi: 10.1136/thoraxjnl-2015-207379. Epub 2015 Oct 26. PMID 26504195
- [Background] Fenger RV, Gonzalez-Quintela A, Vidal C, Husemoen LL, Skaaby T, Thuesen BH, Aadahl M, Madsen F, Linneberg A. The longitudinal relationship of changes of adiposity to changes in pulmonary function and risk of asthma in a general adult population. BMC Pulm Med. 2014 Dec 22;14:208. doi: 10.1186/1471-2466-14-208. PMID 25532602
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Singh SJ, Puhan MA, Andrianopoulos V, Hernandes NA, Mitchell KE, Hill CJ, Lee AL, Camillo CA, Troosters T, Spruit MA, Carlin BW, Wanger J, Pepin V, Saey D, Pitta F, Kaminsky DA, McCormack MC, MacIntyre N, Culver BH, Sciurba FC, Revill SM, Delafosse V, Holland AE. An official systematic review of the European Respiratory Society/American Thoracic Society: measurement properties of field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1447-78. doi: 10.1183/09031936.00150414. Epub 2014 Oct 30. PMID 25359356
- [Background] Eakin EG, Resnikoff PM, Prewitt LM, Ries AL, Kaplan RM. Validation of a new dyspnea measure: the UCSD Shortness of Breath Questionnaire. University of California, San Diego. Chest. 1998 Mar;113(3):619-24. doi: 10.1378/chest.113.3.619. PMID 9515834
- [Background] Mahler DA, Wells CK. Evaluation of clinical methods for rating dyspnea. Chest. 1988 Mar;93(3):580-6. doi: 10.1378/chest.93.3.580. PMID 3342669
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Chai-Coetzer CL, Antic NA, Rowland LS, Catcheside PG, Esterman A, Reed RL, Williams H, Dunn S, McEvoy RD. A simplified model of screening questionnaire and home monitoring for obstructive sleep apnoea in primary care. Thorax. 2011 Mar;66(3):213-9. doi: 10.1136/thx.2010.152801. Epub 2011 Jan 20. PMID 21252389
- [Background] Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009 Oct;124(4):719-23.e1. doi: 10.1016/j.jaci.2009.06.053. Epub 2009 Sep 19. PMID 19767070
- [Background] Schatz M, Sorkness CA, Li JT, Marcus P, Murray JJ, Nathan RA, Kosinski M, Pendergraft TB, Jhingran P. Asthma Control Test: reliability, validity, and responsiveness in patients not previously followed by asthma specialists. J Allergy Clin Immunol. 2006 Mar;117(3):549-56. doi: 10.1016/j.jaci.2006.01.011. PMID 16522452
- [Background] Juniper EF, Guyatt GH, Epstein RS, Ferrie PJ, Jaeschke R, Hiller TK. Evaluation of impairment of health related quality of life in asthma: development of a questionnaire for use in clinical trials. Thorax. 1992 Feb;47(2):76-83. doi: 10.1136/thx.47.2.76. PMID 1549827
- [Background] Juniper EF, Guyatt GH, Willan A, Griffith LE. Determining a minimal important change in a disease-specific Quality of Life Questionnaire. J Clin Epidemiol. 1994 Jan;47(1):81-7. doi: 10.1016/0895-4356(94)90036-1. PMID 8283197
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Juniper EF, Bousquet J, Abetz L, Bateman ED; GOAL Committee. Identifying 'well-controlled' and 'not well-controlled' asthma using the Asthma Control Questionnaire. Respir Med. 2006 Apr;100(4):616-21. doi: 10.1016/j.rmed.2005.08.012. Epub 2005 Oct 13. PMID 16226443
- [Background] Cooper BG. An update on contraindications for lung function testing. Thorax. 2011 Aug;66(8):714-23. doi: 10.1136/thx.2010.139881. Epub 2010 Jul 29. PMID 20671309